CLINICAL TRIAL: NCT03497273
Title: An Open-Label Single-Arm Phase 1 Study Evaluating Safety of Itacitinib in Combination With Corticosteroids for the Treatment of Steroid-Naive Acute Graft-Versus-Host Disease in Japanese Subjects
Brief Title: Safety of Itacitinib in Combination With Corticosteroids for Treatment of Steroid-Naive Acute Graft-Versus-Host Disease in Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 39110-118
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Acute Graft-versus-host Disease
Keywords: JAK1 inhibitor; GVHD; acute GVHD; Japan; corticosteroids
MeSH Terms: interventions — itacitinib; INCB039110; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Itacitinib + corticosteroids (Experimental): Itacitinib administered in combination with corticosteroids.
  Interventions: Drug: Itacitinib; Drug: Corticosteroid

INTERVENTIONS:
Drug: Itacitinib — Itacitinib administered orally once daily at the protocol-defined dose.
  Other Names: INCB039110
Drug: Corticosteroid — Either oral prednisolone or intravenous methylprednisolone at the investigator's discretion.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of itacitinib in combination with corticosteroids in Japanese subjects with Grades II to IV acute graft-versus-host disease (aGVHD).

ELIGIBILITY:
Inclusion Criteria:

* Japanese; subject was born in Japan and has not lived outside of Japan for a total of > 10 years, and subject can trace maternal and paternal Japanese ancestry.
* Has undergone 1 allo-hematopoietic stem cell transplant (HSCT) from any donor and source (unrelated, sibling, haploidentical donors with any matching) using bone marrow, peripheral blood or cord blood for hematologic malignancies. Recipients of myeloablative and reduced-intensity conditioning regimens are eligible.
* Clinically suspected Grades II to IV aGVHD as per Mount Sinai Acute GVHD International Consortium (MAGIC) criteria, occurring after allo-HSCT and any anti-GVHD prophylactic medication.
* Evidence of myeloid engraftment (eg, absolute neutrophil count [ANC] ≥ 0.5 × 10^9/L for 3 consecutive assessments if ablative therapy was previously used). Use of growth factor supplementation is allowed.
* Female subjects should agree to use medically acceptable contraceptive measures, should not be breastfeeding, and must have a negative pregnancy test before the start of study drug administration if of childbearing potential or must have evidence of non-childbearing potential by fulfilling protocol-defined criteria at screening.

Exclusion Criteria:

* Has received more than 1 allo-HSCT.
* Has received more than 2 days of systemic corticosteroids for aGVHD.
* Presence of GVHD overlap syndrome.
* Presence of an active uncontrolled infection (defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs, or radiographic findings attributable to infection; persisting fever without signs or symptoms will not be interpreted as an active uncontrolled infection).
* Known human immunodeficiency virus infection.
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection that requires treatment or at risk for HBV reactivation. For subjects with negative HBsAg and positive total hepatitis B core antibody and for subjects who are positive for HCV antibody, HBV DNA and HCV RNA must be undetectable upon testing.
* Evidence of relapsed primary disease or having been treated for relapse after the allo-HSCT was performed.
* Any corticosteroid therapy (for indication other than GVHD) at doses > 1 mg/kg per day methylprednisolone or equivalent within 7 days of enrollment.
* Severe organ dysfunction unrelated to underlying GVHD, including the following:

  * Cholestatic disorders or unresolved veno-occlusive disease of the liver.
  * Clinically significant or uncontrolled cardiac disease.
  * Clinically significant respiratory disease that requires mechanical ventilation support or 50% oxygen.
* Serum creatinine > 2.0 mg/dL or creatinine clearance < 40 mL/min measured or calculated by Cockroft-Gault equation
* Received Janus kinase (JAK) inhibitor therapy after allo-HSCT for any indication. Treatment with a JAK inhibitor before allo-HSCT is permitted.
* Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | Up to approximately 12 months
  Defined as any adverse event reported for the first time or worsening of a pre-existing event after first dose of study drug.

SECONDARY OUTCOMES:
Cmax of INCB039110 | Up to approximately 1 month
  Maximum observed plasma concentration.
Cl/F of INCB039110 | Up to approximately 1 month
  Apparent oral dose clearance.
Objective response rate | Up to 100 days
  Defined as the proportion of participants demonstrating a complete response, very good partial response, or partial response.
Nonrelapse mortality | Up to approximately 12 months
  Defined as the proportion of participants who died due to causes other than malignancy.
Duration of response | Up to approximately 12 months
  Defined as the interval from first response until GVHD progression or death.
Time to response | Up to approximately 12 months
  Defined as the interval from treatment initiation to first response.
Malignancy relapse rate | Up to approximately 12 months
  Defined as the proportion of participants whose underlying malignancy relapses.
Failure-free survival | Up to 6 months
  Defined as the proportion of participants who are still alive, have not relapsed, have not required additional therapy for aGVHD, and have not demonstrated signs or symptoms of chronic GVHD (cGVHD).
Overall survival | Up to approximately 12 months
  Defined as the interval from study enrollment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Morariu-Zamfir, MD, Study Director — Incyte Corporation
Locations (17):
- Japan (17):
  - JA-Aichi Anjo Kosei Hospital, Anjo-Shi, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hokuyukai Sapporo Hokuyu Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo College of Medicine Hospital, Nishinomiya-Shi, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Jiaikai Imamura General Hospital, Kagoshima, Kagoshima-ken
  - Tokai University Hospital, Isehara-Shi, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - NHO Kumamoto Medical Center, Kumamoto, Kumamoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka City University Hospital, Osaka, Osaka
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - St. Luke's International Hospital, Chūōku, Tokyo-To
  - Jikei University Hospital, Minatoku, Tokyo-To

IPD SHARING:
Plan to Share IPD: No